CLINICAL TRIAL: NCT05204862
Title: A Phase 1/2 Study to Assess Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of TU2218, an Oral TGFβR Inhibitor, Administered Alone and in Combination With Pembrolizumab in Patients With Advanced Solid Tumors
Brief Title: Phase 1/2 Study of TU2218 Alone and in Combination With Checkpoint Inhibitors in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TiumBio Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TUC1PI-01
Record Dates: First submitted 2021-12-21; First posted 2022-01-24 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — spartalizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- TU2218 Phase 1a (Experimental): Escalating doses of TU2218 orally administered daily for two weeks followed by one week of rest for up to 21-day cycles
  Interventions: Drug: TU2218
- TU2218 Food Effect (Experimental): TU2218 orally administered at a one dose level below MTD under fasting condition on -Day 2, followed by the same dose orally administered with meals on -Day 1 and then continued under fasted condition for two weeks followed by one week of rest for up to 21-day cycles
  Interventions: Drug: TU2218
- TU2218 + Anti-PD-1 antibody Phase 1b (Experimental): Escalating doses of TU2218 in combination with anti-PD-1 antibody up to 21-day cycles
  Interventions: Drug: TU2218; Drug: Anti-PD-1 antibody
- TU2218 Phase 2a (Experimental): TU2218 at a RP2D orally administered daily for two weeks followed by on week of rest for up to 21-day cycles
  Interventions: Drug: TU2218
- TU2218 + Anti-PD-1 antibody Phase 2b (Experimental): TU2218 at a RP2DC in combination with anti-PD-1 antibody up to 21-day cycles
  Interventions: Drug: TU2218; Drug: Anti-PD-1 antibody

INTERVENTIONS:
Drug: TU2218 — orally administered
Drug: Anti-PD-1 antibody — Intravenously administered
  Arms: TU2218 + Anti-PD-1 antibody Phase 1b; TU2218 + Anti-PD-1 antibody Phase 2b

SUMMARY:
This study consists of Part A for monotherapy and Part B for combination therapy to evaluate safety, tolerability, pharmacokinetics, and preliminary efficacy of TU2218 in patients with advanced solid tumors. The main purpose of Phase 1 is to determined the recommended Phase 2 dose (RP2D) of TU2218 and the main purpose of Phase 2 is to evaluate the antitumor activity of TU2218 at RP2D.

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least 18 years of age at the time of consent (ie, screening), or according to local regulatory requirement if the legal age for consenting for study participation is more than 18 years.
* Life expectancy ≥12 weeks as judged by the Investigator.
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1; except for Phase1a that can enroll patients with either measurable and/or non-measurable disease.
* Eastern Cooperative Oncology Group (ECOG) 0 or 1.
* Able to swallow capsules.
* Histologically or cytologically documented advanced solid tumor for which no effective standard therapy exists, or standard therapy has failed (Phase 1a).
* Histologically or cytologically documented advanced solid tumor for which no effective standard therapy exists, and for which standard therapy containing an anti-PD-(L)1 agent has failed after an initial response or stabilization of at least 4-month duration (Phase 1b and 2a).
* Adequate hematological function, coagulation defined by:

  1. Absolute neutrophil count ≥1,500 cells/μL
  2. Platelet count ≥100,000/μL
  3. Hemoglobin ≥9.0 g/dL
  4. International normalized ratio <1.5 × the upper limit of normal (ULN)
* Adequate hepatic and renal functions defined by:

  1. Total bilirubin ≤1.5 × ULN
  2. AST and ALT ≤3 × ULN; if liver metastases are present, then ≤5 × ULN is allowed
  3. Estimated creatinine clearance >60 mL/min according to the Cockcroft-Gault formula
* Able to understand and to comply with all protocol requirements, instructions, and restrictions.
* QT interval corrected using Fridericia's formula (QTcF) interval ≤460 msec on screening ECG.
* Normal ejection fraction (within the reference range of the institution).
* A washout period of 4 weeks for any biologic material and a minimum of 5 half-lives for any chemotherapy is required prior to the start of treatment with resolution of any toxicity to maximum Grade 1 (except alopecia)
* Completion of radiotherapy at least 14 days prior to the start of treatment with resolution of any toxicity to maximum Grade 1
* Female patients of childbearing potential must have a negative serum pregnancy test within 7 days of the first administration of study treatment. For the purpose of this study, female patients of childbearing potential are defined as all female after puberty unless they are postmenopausal for at least 1 year, or are surgically sterile (hysterectomy or bilateral oophorectomy or tubal ligation)

Exclusion Criteria:

* Myocardial infarction within 6 months prior to screening, or pericardial effusion.
* History of cardiac or aortic surgery within 6 months prior to screening.
* Unstable angina pectoris, cerebrovascular accident, transient ischemic attack, or symptomatic pulmonary embolism; deep venous thrombosis; arterial occlusive disease in the past 12 months.
* Congestive heart failure of New York Heart Association class III/IV.
* Major arrhythmia or abnormalities identified by ECG per Investigator's judgment.
* Uncontrolled hypertension (as defined by systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg) during the screening period.
* Elevated troponin 1 levels (Grade 3) at screening or known to have persistently elevated brain natriuretic peptide.
* Active and clinically significant bacterial, fungal, or viral infection, including active or known history of hepatitis B virus (defined as hepatitis B surface antigen [HbsAg] reactive), or known active hepatitis C virus (defined as hepatitis C virus ribonucleic acid [qualitative] is detected), known human immunodeficiency virus or acquired immunodeficiency syndrome related illness. However, an inactive hepatitis B virus carrier can be enrolled
* Current or history of interstitial pneumonitis.
* Uncontrolled metastatic disease to the brain or central nervous system, massive uncontrolled effusions (pleural, pericardial, peritoneal), pulmonary lymphangitis, and over 50% liver involvement that is at the discretion of the Investigator. Note: Pleural effusion should be defined by Investigator's discretion.
* Known history of difficulty swallowing, malabsorption or other conditions that may reduce absorption of the product.
* Received prior treatment targeting the signaling pathway of TGF-β.
* Tumor that compresses or invades major blood vessels or tumor cavitation that in the opinion of the Investigator is likely to bleed.
* History of severe bleeding. Unable to stop anticoagulation therapy with heparin, low molecular weight heparin, vitamin K antagonists, antiplatelet agents, or factor Xa inhibitors throughout the study and for at least 28 days after the last administration of study treatment.
* Regular use of aspirin (>325mg/day) or other non-steroidal anti-inflammatory drugs with antiplatelet activity or treatment with dipyramidole, ticlopidine, clopidogrel, or cilostazol within 10 days of first administration of study treatment.
* Moderate or severe heart valve function defect including moderate or severe valve stenosis or regurgitation.
* Evidence or history of septal aneurysm, other heart aneurysm, or any aneurysm of the major vessels.
* Active infection requiring systemic antibiotic therapy.
* Receipt of any live vaccine or live-attenuated vaccine within 30 days prior to the first drug administration and while participating the study.
* Unable to unwilling to stop use of strong inhibitors of CYP1A2, CYP2C8, and CYP3A4, and strong inhibitors of P-gp and BCRP at least 8 days prior to study entry (Day 1) or within all dose escalation cohorts.
* Unable or unwilling to stop use of gastric pH elevating agents including proton pump inhibitors, H2-recpetor antagonists and antacide at least 8 days prior to study entry (Day 1) or within all dose escalation cohorts.
* Unwilling to stop use of herbal supplements or traditional herbal medicines.
* Known substance abuse concurrent treatment with non-permitted drugs.
* Known history, or suspected hypersensitivity to any excipients of the clinical study drugs.
* Undergone major surgeries within 28 days of first dosing, or have a planned surgery during the study period.
* Female patients who are breastfeeding.
* Female patients must not be pregnant or at risk to become pregnant during the study. Fertile male and female patients must agree to use an effective barrier method of birth control to avoid pregnancy (for female patients a double-barrier method of contraception, for male patients a condom with spermicide) or total abstinence from the time of providing informed consent until 30 days after the last administration of TU2218.
* Any other serious medical condition which in the Investigator's opinion would preclude safe participation in the study.

For Anti PD1 antibody combination therapy part:

* Unable to stop chronic systemic steroid therapy or any other immunosuppressive mediacation
* Use of oral, inhaled, or topical corticosteroid, at doses > 10mg/day prednisolone or equivalent and the dose must be stable over 4 weeks prior to Day1 of Cycle1.
* Active autoimmune disease or history of autoimmune disease, except vitiligo, hypothyroidism, or resolved childhood asthma/atropy
* Known tolerance to an anti-PD(L)1 agent during prior exposure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-12-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Maximum Tolerated Dose (MTD) of TU2218 administered alone (Part A) and in combination with anti-PD-1 antibody (Part B) | From the beginning of Cycle 1 through Cycle 2 (each cycle is 21 days)
  The MTD is determined as DLTs.
Phase 2: Overall Response rate (ORR) of TU2218 administered alone (Part A) and in combination with anti-PD-1 antibody (Part B) | 24 weeks
  ORR is defined as the proportion of patients who have a PR and CR.

SECONDARY OUTCOMES:
Incidence of treatment-emergent AEs | approximately 13 months
  TEAE is defined as treatment-emergent changes in clinical laboratory values, ECG, vital signs, ECOG performance scores, and physical examination findings.
Peak Plasma Concentration (Cmax) of TU2218 for TU2218 alone and in combination with anti-PD1 antibody | Cycle 1
  Cmax is defined as the maximum observed concentration of the drug in plasma.
Area under the plasma concentration versus time curve (AUC) of TU2218 for TU2218 alone and in combination with anti-PD1 antibody | Cycle 1
  AUC is defined as the definite integral of a curve that describes the variation of a drug concentration in plasma as a function of time.
Terminal half-life (t1/2) of TU2218 for TU2218 alone and in combination with anti-PD1 antibody | Cycle 1
  Half-life is defined as the time required to divide the plasma concentration by two after reaching pseudo-equilibrium.
Clearance (CL) of TU2218 for TU2218 alone and in combination with anti-PD1 antibody | Cycle 1
  CL is defined as the volume of plasma from which a substance is completely removed per unit time.
Duration of Response (DoR) | over 24 weeks
  DoR is measured from the date of documented response to the date of first progression of disease or the date of death due to any cause, whichever is earlier.
Progression Free Survival (PFS) | over 24 weeks
  PFS is defined as the time from the date of first study treatment to the first evidence of disease progression as defined by response evaluation criteria in solid tumors (RECIST) v1.1 or iRECIST.
Overall Survival (OS) | Date of First Study Treatment to Death from Any Cause (up to 24 months)
  OS is determined from the date of first study treatment until death due to any cause.
Clinical benefit rate (CBR) | over 24 weeks
  CBR is defined as the proportion of patients with the best overall response as CR, PR or SD (lasting at least 24 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: TU2218, Study Director — TiumBio Co., Ltd.
Locations (3):
- NEXT Oncology, San Antonio, Texas, United States
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No
We will make our final decision after EOP2 meeting.